CLINICAL TRIAL: NCT02198976
Title: Australian Barrett's Cohort With Dysplasia and Early Cancer Study
Acronym: ABCDE
Status: Recruiting | Type: Observational
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Other Study IDs: HREC2013/10/4.1 (3829)
Record Dates: First submitted 2014-07-17; First posted 2014-07-24 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Barrett's Oesophagus: Patients with Barrett's Oesophagus with either high grade dysplasia (HGD) or intramucosal cancer (IMC)

SUMMARY:
The purpose of this study is to collect prospective observational data regarding endoscopic management and outcomes of patients with Barrett's oesophagus (BO) with high grade dysplasia and/or intramucosal carcinoma. To observe the natural history of patients with low grade dysplastic and non dysplastic Barrett's oesophagus

ELIGIBILITY:
Inclusion Criteria:

* Can give informed consent to trial participation
* Age greater than 18
* Barrett's oesophagus

Exclusion Criteria:

* Age less than 18
* Pregnant patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient's presenting to tertiary referral study site with HGD or IMC Barrett's Oesophagus for removal.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-04; Primary Completion 2034-05 (Estimated); Study Completion 2034-11 (Estimated)

PRIMARY OUTCOMES:
Number of Serious and Non-Serious Adverse Events | During the Barretts Excision
  Collect prospective observational data on patients undergoing endoluminal therapy for dysplastic BO to determine
  * Long term risk of oesophageal adenocarcinoma (OAC) development
  * Long term efficacy (dysplasia and metaplasia free) in both long and short segment BO
  * Short and long term safety and complications
  * Comparison of the safety, long term efficacy, cost and patient tolerability between endoscopic mucosal resection (EMR) and radiofrequency ablation (RFA) Document the endoscopic location and characterise morphology of HGD/IMC in short and long segment BO Define the short term and long term causes of morbidity / mortality of patients undergoing ER This will be recorded on a datasheet, de-identified during the procedure.

SECONDARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | Up to 5 years after procedure
  Establish the effect of endoluminal therapies for BO HGD/IMC on oesophageal motility. Document and grade the post EMR oesophageal defect and establish a possible link to subsequent complications (including stricture, bleeding and perforation) and recurrence. Perform cost-utility analyses comparing different treatment approaches for BO HGD/IMC, including EMR, RFA and oesophagectomy. Establish the relationship between Obstructive Sleep Apnea and BO. Understand patient attitudes and perceptions regarding BO, its treatment and its implication.
  Participants will be approached following their procedure and data recorded on a datasheet, this data will be linked to the initial procedure outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bourke, MBBS, Principal Investigator — Western Sydney Local Health District
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia